CLINICAL TRIAL: NCT02053571
Title: Evaluation of 3D Overlay During Transjugular Intrahepatic Portosystemic Shunt (TIPS) Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Siemens Medical Solutions (Industry)
Responsible Party: Principal Investigator, Robert A. Hieb, MD, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO19417
Record Dates: First submitted 2014-01-24; First posted 2014-02-03 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Portal Hypertension
MeSH Terms: conditions — Hypertension, Portal | interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TIPS with 3D overlay (Experimental)
  Interventions: Procedure: TIPS with 3D Overlay

INTERVENTIONS:
Procedure: TIPS with 3D Overlay

SUMMARY:
The goal of this study is to evaluate an alternate approach, which involves using a 3D puncture path overlay, to access the portal vein during a Transjugular Intrahepatic Portosystemic Shunt (TIPS) procedure. The study should determine if the alternate approach provides these benefits: improved safety of procedure, and reduced intervention time (including reduction of radiation exposure), which benefits both interventional radiologist and the patient.

During a TIPS procedure, a shunt or stent (mesh tube) is passed down the jugular vein (the vein above the collarbone in the neck) using fluoroscopy (x-ray) guidance. The shunt then is inserted between the portal vein (vein that carries blood from the digestive organs into the liver) to a hepatic vein (vein that carries blood away from the liver back to the heart).

In the standard approach, the interventional radiologist uses two-dimensional guidance (2D - having the dimensions of height and width only) to locate the path between the portal vein and hepatic vein. However, since these two veins do not connect, this method does not provide information on the three-dimensional (3D) relationship between the two veins.

In the alternate approach, the physician will have the option of using 3D guidance to locate the path. An on-table limited (small field of view) CT scan, used in combination with FDA approved imaging software, will provide a 3D image demonstrating the relationship between the portal vein and the hepatic vein. The 3D image is overlaid on the standard live x-ray images to assist in needle guidance during the TIPS procedure.

The CT scan performed will be in place of the angiograms that are typically performed. However, if the portal vein is not adequately seen in the CT images, the angiograms will be done and there will be no overlay. The procedure will proceed using the standard approach.

ELIGIBILITY:
Inclusion Criteria:

* Prospective study of 20 patients, age 18 years or older, scheduled for clinically indicated TIPS procedure. Patients must be capable of providing informed consent.

Exclusion Criteria:

* does not meet inclusion criteria.
* portal vein does not opacify

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-04; Primary Completion 2016-08-04 (Actual); Study Completion 2016-08-04 (Actual)

PRIMARY OUTCOMES:
The number of cases in which the portal vein anatomy is accurately delineated in 3D using this technique | At time of procedure

SECONDARY OUTCOMES:
x-ray dose | At time of procedure
Procedure time | At time of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Hieb, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin/Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No